CLINICAL TRIAL: NCT07377344
Title: Closing Health Equity Through Empowering Oral Health for Maternal Wellness
Brief Title: CHEER Oral Health in Pregnancy Study
Acronym: CHEER
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Colgate Palmolive (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20254330
Record Dates: First submitted 2026-01-12; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Gingivitis; Dental Health; Pregnancy; Pregnancy Outcomes; Randomized Controlled Trial; Periodontal Disease; Gum Disease
MeSH Terms: conditions — Gingivitis; Periodontal Diseases; Gingival Diseases

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test (Experimental): Enhanced Care + receive a home oral care kit (toothbrush, toothpaste, and floss), structured oral hygiene education, and behavioral reinforcement via weekly surveys
  Interventions: Behavioral: Enhanced Care +
- Control (Other): Participants receive "enhanced care" where they received standard oral hygiene education at the baseline visit. Do NOT receive oral care kit (toothbrush, toothpaste, and floss), structured oral hygiene education, and behavioral reinforcement via weekly surveys
  Interventions: Behavioral: Enhanced Care

INTERVENTIONS:
Behavioral: Enhanced Care — All participants receive standard oral hygiene education at the baseline visit.
  Arms: Control
Behavioral: Enhanced Care + — All participants receive standard oral hygiene education at the baseline visit. Test participants also receive a home oral care kit (toothbrush, toothpaste, and floss), and will start receiving weekly oral health check-ins and reminder surveys following their initial visits at one-week intervals starting the day after their baseline visit
  Arms: Test

SUMMARY:
Many pregnant people don't get the dental care they need, even though it's safe and important. The CHEER Study offers free dental check-ups, cleanings, and supplies to help participants take care of their teeth and gums during pregnancy. The purpose of this research study is to compare two types of noninvasive oral health interventions to evaluate their effectiveness. We want to learn if one method is more effective in supporting oral health and improving pregnancy outcomes. There are two aims of this study:

Aim 1: To evaluate whether a structured oral health intervention reduces periodontal inflammation during pregnancy and postpartum in pregnant people with indicators of periodontal disease.

Aim 2: To assess whether a structured oral health intervention is associated with changes in oral health behaviors or birth outcomes in pregnant people with periodontal disease.

DETAILED DESCRIPTION:
The Closing Health Equity through Empowering Oral Health for Maternal Wellness (the CHEER Oral Health in Pregnancy Study) aims to address significant oral health disparities experienced by pregnant individuals, particularly those from low-income and minority communities in California.

Oral health is a critical yet often overlooked component of prenatal care. Existing evidence suggests that periodontal disease is associated with adverse pregnancy outcomes, such as preterm birth and low birth weight. However, many pregnant individuals in California do not receive adequate oral health services, especially those from historically marginalized communities. The CHEER Project aims to address this gap by implementing an intervention that is scalable, community-engaged, and grounded in evidence-based education.

This study will generate novel data on the impact of oral health education and behavior modification, delivered through accessible messaging and product use, on periodontal inflammation and disease status, and microbiome profiles. It will also explore potential downstream effects on perinatal outcomes. The study aligns with public health priorities to improve maternal wellness, health equity, and the integration of dental and medical care.

There are two study aims:

Aim 1: To evaluate whether a structured oral health intervention reduces periodontal inflammation during pregnancy and postpartum in pregnant people with indicators of periodontal disease.

Aim 2: To assess whether a structured oral health intervention is associated with changes in oral health behaviors or birth outcomes in pregnant people with periodontal disease.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant individuals aged 18 years or older with indications of periodontal diseases (gingivitis or mild periodontitis, moderate to severe periodontitis)
2. Less than 20 weeks pregnancy at time of enrollment
3. Has dental insurance (Medi-Cal or private coverage)
4. Willing and able to provide informed consent
5. Planning to receive ongoing prenatal care at study-affiliated clinics
6. Access to a mobile phone for receiving text messages

Exclusion Criteria:

1. Presence of systemic diseases or medical conditions that require antibiotic prophylaxis for dental procedures
2. Current immunosuppressive therapy/use of anti-inflammatory medications
3. Receipt of active periodontal treatment within the past 6 months
4. Complete edentulism (no natural teeth)
5. Unable to read and write English
6. Less than 9th grade education
7. Enrollment in another oral interventional study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2028-02-01 (Estimated); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
Change in periodontal inflammation | 28 weeks
  Change in periodontal inflammation by survey and exam from baseline to 28-<36 weeks gestation to postpartum follow-up.

SECONDARY OUTCOMES:
Changes in oral health behaviors | 28 weeks
  Change in patient reported 1) teeth brushing twice a day, 2) teeth brushing for two minutes each time, 3) daily use of floss among test and control participants
Difference in birth outcomes between test and control groups | 28 weeks
  Differences between test and control participants: total weeks gestational age at delivery, preterm birth (<37 gestational weeks), birthweight (in grams), low birth weight delivery (<2500 grams), growth for gestational age percentile, and small for gestational age infant (infant birth weight lower than 10th percentile).

CONTACTS AND LOCATIONS:
Overall Officials: Effie Ioannidou, DDS, MDS, Principal Investigator — University of California, San Francisco; Laura Jelliffe-Pawlowski, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Dental Center, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No